CLINICAL TRIAL: NCT06956833
Title: Self-Guided Versus Facilitator-Guided Debriefing in Immersive Virtual Reality Simulation: Protocol for a Randomized Controlled Non-Inferiority Trial As-sessing Teamwork Skills in Medical Students
Brief Title: Immersive Virtual Reality Simulation-Effects of Self-Guided Versus Facilitator-Guided Debriefing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Amalie Middelboe Andersen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: P-2023-167
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Virtual Reality Simulation; Simulation-based Medical Education; Pediatric Emergency Medicine; Immersive Virtual Reality; Debriefing
Keywords: Immersive Virtual Reality; Virtual Reality simulation; Simulation-based medical education; Pediatric emergencies; Debriefing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-guided debriefing (Experimental): Immersive virtual reality simulation-based pediatric emergency training with self-guided debriefing
  Interventions: Other: Ìmmersive virtual reality simulation with self-guided debriefing
- Facilitator-guided debriefing (Active Comparator): Immersive virtual reality simulation-based pediatric emergency training with facilitator-guided debriefing
  Interventions: Other: Ìmmersive virtual reality simulation with facilitator-guided debriefing

INTERVENTIONS:
Other: Ìmmersive virtual reality simulation with self-guided debriefing — * Familiarization with immersive virtual reality simulation (1 hour)
  * Video tutorial introducing paediatric Airway, Breathing, Circulation, Disability, Exposure (ABCDE) assessment, emergency teamwork and communication, and core elements in debriefing (1 hour)
  * Three immersive virtual reality simulation-based pediatric emergency team training scenarios with self-guided debriefing (2 hours)
  Arms: Self-guided debriefing
Other: Ìmmersive virtual reality simulation with facilitator-guided debriefing — * Familiarization with immersive virtual reality simulation (1 hour)
  * Video tutorial introducing paediatric ABCDE assessment, emergency teamwork and communication, and core elements in debriefing (1 hour)
  * Three immersive virtual reality simulation-based pediatric emergency team training scenarios with facilitator-guided debriefing (2 hours)
  Arms: Facilitator-guided debriefing

SUMMARY:
The goal of this clinical trial is to find out whether self-guided and facilitator-guided virtual reality (VR) simulations are equally effective in helping medical students learn how to manage and treat critically ill children. The study will also investigate how medical students feel about the two training methods and examine how many experience cybersickness. The main questions it aims to answer are:

* Does self-guided VR simulation work as well as facilitator-guided VR simulation in teaching medical students how to manage critically ill children?
* How do medical students experience the ease of use, workload, reflection on learning, and motivation in each training method?
* How many students experience cybersickness? To answer these questions, researchers will compare the two training methods to evaluate if self-guided VR simulation is an effective way to teach medical students how to manage critically ill children.

Participants will:

* Work through three VR cases to practice managing critically ill children in a safe environment.
* Be tested before and after the VR simulation to assess changes in their skills managing critically ill children.
* Complete surveys about their experience of the VR simulation, the training sessions, and any cybersickness symptoms they might have.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be medical students enrolled at medical schools in Denmark who are within two years of graduation.

Exclusion Criteria:

* Lack of informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Clinical Teamwork Scale | The medical students will be videorecorded at Day 1 (intervention day) immediately before and after the intervention. Two raters will assess the videos once all data collection for the trial has been completed.
  The investigators will assess medical students' teamwork skills using the Clinical Teamwork Scale (CTS). This validated scale assesses fifteen teamwork skills across five main domains: overall teamwork, communication, situational awareness, decision-making, and role responsibility, on an 11-point Likert scale ranging from 1 = unacceptable to 11 = perfect. The CTS has been translated into Danish using a forward-backward translation process by two professional translators.
  Medical students will be videorecorded immediately before and after the intervention while managing a mannequin-based pediatric emergency in teams of two. Two independent raters will assess each team's collective performance based on the videos, using the CTS.

SECONDARY OUTCOMES:
ABCDE checklist | The medical students will be videorecorded at Day 1 (intervention day) immediately before and after the intervention. Two raters will assess the videos once all data collection for the trial has been completed.
  The investigators will assess medical students' adherence to the Airways, Breathing, Circulation, Disability, Exposure (ABCDE) approach using the ABCDE checklist. Modified from an ABCDE checklist for adult life support, this checklist assesses adherence to the European Paediatric Advanced Life Support guidelines for ABCDE assessment and ranges from 0 = not initiated to 3 = performed consistently during the whole simulation.
  Medical students will be videorecorded immediately before and after the intervention while managing a mannequin-based pediatric emergency in teams of two. Two independent raters blinded to group allocation will assess each team's collective performance based on the videos, using the ABCDE checklist.
Time to critical action | The medical students will be videorecorded at Day 1 (intervention day) immediately before and after the intervention. Two raters will assess the videos once all data collection for the trial has been completed.
  The investigators will assess medical students' time to critical actions measured as time in seconds to administration of oxygen (pneumonia case) or beta2 agonist (asthma case), administration of a fluid bolus (10 mL/kg body weight), and completion of the ABCDE assessment. If the team does not perform the action, they will be assigned a time of 900 seconds.
  Medical students will be video recorded before and after the intervention while managing a mannequin-based pediatric emergency in teams of two. Two independent raters blinded to group allocation will assess each team's time to predefined critical actions based on the videos.
Debriefing Assessment for Simulation in Healthcare Student Version | Medical students will complete the DASH-SV questionnaire at Day 1 (the intervention day) after each debriefing.
  This validated questionnaire is designed for learners to evaluate a debriefing on a 7-point Likert scale ranging from 1 = extremely ineffective to 7 = extremely effective. In consultation with the Debriefing Assessment for Simulation in Healthcare Student Version (DASH-SV©) developers, the investigators have replaced 'The facilitator' with 'We' in the self-guided debriefing group to fit the context. DASH-SV has been translated into Danish using a forward-backward translation process by two professional translators.
Intrinsic Motivation Inventory | Medical students will complete the IMI questionnaire at Day 1 (intervention day) after completion of the intervention.
  This validated questionnaire measures the subjective motivation related to a specific activity on a 7-point Likert scale ranging from 1 = not at all true to 7 = very true. Intrinsic Motivation Inventory (IMI) consists of 22 items across four domains: interest/enjoyment (seven items), perceived competence (five items), perceived choice (five items), and pressure/tension (five items). In this study, the investigatorswill use the seven-item Interest/Enjoyment domain, which is considered the direct measure of intrinsic motivation. IMI has previously been translated professionally to Danish and tested in a Danish context.
System Usability Scale | Medical students will complete the SUS questionnaire at Day 1 (intervention day) after completion of the intervention.
  This validated questionnaire measures the subjective usability of a product on a 5-point Likert scale ranging from 1 = strongly disagree to 5 = strongly agree. The System Usability Scale (SUS) item scores are subsequently converted into a single SUS score on a scale from 0 to 100 (0 = lowest, 100 = highest). SUS has previously been translated professionally to Danish and validated in a Danish context.
NASA Task Load Index | Medical students will complete the NASA-TLX at Day 1 (intervention day) after completion of the intervention.
  This validated scale measures subjective workload related to a specific activity. The scale ranges from 0 to 21, and the item scores are subsequently converted into a single score from 0 to 100 (0 = lowest, 100 = highest). National Aeronautics and Space Administration Task Load Index (NASA-TLX) has been translated into Danish using a forward-backward translation process by two professional translators.
Virtual Reality Sickness Questionnaire | Medical students will complete the VRSQ questionnaire at Day 1 (intervention day) after completion of the intervention.
  Virtual Reality Sickness Questionnaire(VRSQ) is a validated questionnaire designed to measure symptoms of cybersickness experienced during immersive virtual reality use. It evaluates nine symptoms on a Likert-type scale ranging from 0 = none to 3 = severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooke J. SUS: A 'Quick and Dirty' Usability Scale. In: Jordan PW, Thomas B, Weerdmeester BA, McClelland IL, editors. Usability Evaluation In Industry. London: Taylor & Francis; 1996. p. 189-94.
- [Background] https://doi.org/10.1016/j.apergo.2017.12.016
- [Background] Hart SG, Staveland LE. Development of NASA-TLX (Task Load Index): Results of Empirical and Theoretical Research. Advances in Psychology. 1988 Jan 1;52(C):139-83.
- [Background] Brett-Fleegler M, Rudolph J, Eppich W, Monuteaux M, Fleegler E, Cheng A, Simon R. Debriefing assessment for simulation in healthcare: development and psychometric properties. Simul Healthc. 2012 Oct;7(5):288-94. doi: 10.1097/SIH.0b013e3182620228. PMID 22902606
- [Background] https://doi.org/10.1016/j.resuscitation.2021.02.015
- [Background] Hultin M, Jonsson K, Hargestam M, Lindkvist M, Brulin C. Reliability of instruments that measure situation awareness, team performance and task performance in a simulation setting with medical students. BMJ Open. 2019 Sep 12;9(9):e029412. doi: 10.1136/bmjopen-2019-029412. PMID 31515425
- [Background] Guise JM, Deering SH, Kanki BG, Osterweil P, Li H, Mori M, Lowe NK. Validation of a tool to measure and promote clinical teamwork. Simul Healthc. 2008 Winter;3(4):217-23. doi: 10.1097/SIH.0b013e31816fdd0a. PMID 19088666
- [Background] Abulfaraj MM, Jeffers JM, Tackett S, Chang T. Virtual Reality vs. High-Fidelity Mannequin-Based Simulation: A Pilot Randomized Trial Evaluating Learner Performance. Cureus. 2021 Aug 11;13(8):e17091. doi: 10.7759/cureus.17091. eCollection 2021 Aug. PMID 34527478
- [Background] Umoren R, Bucher S, Hippe DS, Ezenwa BN, Fajolu IB, Okwako FM, Feltner J, Nafula M, Musale A, Olawuyi OA, Adeboboye CO, Asangansi I, Paton C, Purkayastha S, Ezeaka CV, Esamai F. eHBB: a randomised controlled trial of virtual reality or video for neonatal resuscitation refresher training in healthcare workers in resource-scarce settings. BMJ Open. 2021 Aug 25;11(8):e048506. doi: 10.1136/bmjopen-2020-048506. PMID 34433598
- [Background] Farra S, Hodgson E, Miller ET, Timm N, Brady W, Gneuhs M, Ying J, Hausfeld J, Cosgrove E, Simon A, Bottomley M. Effects of Virtual Reality Simulation on Worker Emergency Evacuation of Neonates. Disaster Med Public Health Prep. 2019 Apr;13(2):301-308. doi: 10.1017/dmp.2018.58. Epub 2018 Oct 8. PMID 30293544
- [Background] Zackoff MW, Real FJ, Sahay RD, Fei L, Guiot A, Lehmann C, Tegtmeyer K, Klein M. Impact of an Immersive Virtual Reality Curriculum on Medical Students' Clinical Assessment of Infants With Respiratory Distress. Pediatr Crit Care Med. 2020 May;21(5):477-485. doi: 10.1097/PCC.0000000000002249. PMID 32106189
- [Background] Foronda CL, Gonzalez L, Meese MM, Slamon N, Baluyot M, Lee J, Aebersold M. A Comparison of Virtual Reality to Traditional Simulation in Health Professions Education: A Systematic Review. Simul Healthc. 2024 Jan 1;19(1S):S90-S97. doi: 10.1097/SIH.0000000000000745. Epub 2023 Aug 31. PMID 37651101
- [Background] Cook DA, Hatala R, Brydges R, Zendejas B, Szostek JH, Wang AT, Erwin PJ, Hamstra SJ. Technology-enhanced simulation for health professions education: a systematic review and meta-analysis. JAMA. 2011 Sep 7;306(9):978-88. doi: 10.1001/jama.2011.1234. PMID 21900138
- [Background] Thim S, Henriksen TB, Laursen H, Schram AL, Paltved C, Lindhard MS. Simulation-Based Emergency Team Training in Pediatrics: A Systematic Review. Pediatrics. 2022 Apr 1;149(4):e2021054305. doi: 10.1542/peds.2021-054305. PMID 35237809
- [Derived] Sohlin AM, Poulsen A, Hoffmann IM, Gjaerde LK, Lund S, Overbeck G, Paulsen L, Chang TP, Lee JY, Sorensen JL, Kjaergaard J. Self-guided versus facilitator-guided debriefing in immersive virtual reality simulation: Protocol for a randomized controlled non-inferiority trial assessing teamwork skills in medical students. PLoS One. 2025 Sep 12;20(9):e0332309. doi: 10.1371/journal.pone.0332309. eCollection 2025. PMID 40938855